CLINICAL TRIAL: NCT01129531
Title: A Study of the Safety and Efficacy of AGN-214868 in Patients With Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214868-002
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-09

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AGN-214868 3.25 μg (Experimental): AGN-214868 injected into areas of postherpetic neuralgia pain for a total dose of 3.25 μg per treatment.
  Interventions: Drug: AGN-214868
- AGN-214868 16.25 μg (Experimental): AGN-214868 injected into areas of postherpetic neuralgia pain for a total dose of 16.25 μg per treatment.
  Interventions: Drug: AGN-214868
- Placebo (Placebo Comparator): Placebo to AGN-214868 injected into areas of postherpetic neuralgia pain per treatment.
  Interventions: Drug: Placebo to AGN-214868

INTERVENTIONS:
Drug: AGN-214868 — AGN-214868 injected into areas of postherpetic neuralgia pain for total dose per treatment.
  Arms: AGN-214868 16.25 μg; AGN-214868 3.25 μg
Drug: Placebo to AGN-214868 — Placebo to AGN-214868 injected into areas of postherpetic neuralgia pain per treatment.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of AGN-214868 in patients with postherpetic neuralgia (PHN) - nerve pain.

ELIGIBILITY:
Inclusion Criteria:

* Persistent postherpetic neuralgia (PHN) with nerve pain present for at least 9 months after onset of herpes zoster skin rash

Exclusion Criteria:

* Female patients with reproductive potential
* Active herpes zoster skin rash
* Current or anticipated treatment with acupuncture, TNS, or steroids
* Current or anticipated use of topical analgesic agents with PHN
* Treatment with botulinum toxin therapy of any serotype within the prior 12 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Orlando, Florida, United States
- Brno, Czechia
- Kiel, Kiel, Germany
- Katowice, Poland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were two Treatment Cycles in this study 12 weeks apart. In Treatment Cycle 1 participants were randomized to AGN-214868 3.25 μg, AGN-214868 16.25 μg or Placebo. In Treatment Cycle 2 participants were re-randomized to AGN-214868 3.25 μg, AGN-214868 16.25 μg or Placebo.
Period: Treatment Cycle 1
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Started | 84 | 84 | 126
Completed | 80 | 78 | 110
Not Completed | 4 | 6 | 16
Period: Treatment Cycle 2
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Started | 94 (Participants who completed Treatment Cycle 1 were re-randomized.) | 95 (Participants who completed Treatment Cycle 1 were re-randomized.) | 79 (Participants who completed Treatment Cycle 1 were re-randomized.)
Completed | 88 | 92 | 74
Not Completed | 6 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo | Total
Number analyzed (Participants) | 84 | 84 | 126 | 294
Age, Customized [Number; unit: Participants]
  18 to < 40 Years | 2 | 2 | 2 | 6
  40 to < 65 Years | 18 | 29 | 38 | 85
  65 to < 75 Years | 42 | 33 | 57 | 132
  ≥ 75 Years | 22 | 20 | 29 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 73 | 164
  Male | 40 | 37 | 53 | 130

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Pain Intensity Score at Week 12
Description: Participants rated the severity of their daily pain in the previous 7 days using a 10 point scale where 0=no pain to 10=pain as bad as you can imagine. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Modified intent to treat population included all randomized participants who received treatment and had at least 1 post-baseline pain intensity score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Number analyzed (Participants) | 84 | 82 | 124
Score on a scale
  Baseline | 6.13 (1.248) | 6.04 (1.324) | 6.05 (1.334)
  Change from Baseline at Week 12 | -1.42 (1.876) | -1.35 (1.996) | -1.27 (2.036)

2. Secondary Outcome: Change From Baseline in Area of Spontaneous Pain
Description: A tracing of the area of spontaneous pain was made and sent to an independent central reading center for measurement. The area of spontaneous pain was measured in centimeters squared (cm^2) at Baseline and Week 12. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Number analyzed (Participants) | 84 | 82 | 124
cm^2
  Baseline | 87.44 (51.312) | 118.17 (74.858) | 98.27 (62.866)
  Change from Baseline at Week 12 (N=81, 79, 117) | -4.83 (62.374) | -17.18 (62.694) | -6.13 (68.990)

3. Secondary Outcome: Change From Baseline in Area of Allodynia
Description: A tracing of the area of allodynia (pain to touch) was made and sent to an independent central reading center for measurement. The area of allodynia was measured in centimeters squared (cm^2) at Baseline and Week 12. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- Placebo: Placebo to AGN-214868 injected into areas of postherpetic neuralgia pain per treatment. Participants received two treatments 12 weeks apart.
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Number analyzed (Participants) | 84 | 82 | 124
cm^2
  Baseline | 184.28 (145.259) | 195.11 (149.355) | 174.17 (134.132)
  Change from Baseline at Week 12 (N=81, 79, 117) | -32.40 (89.849) | -43.56 (107.183) | -15.27 (116.338)

4. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia
Description: Participants were asked to rate the unpleasantness (pain to touch) after 3 brush strokes in the area of allodynia on a 100 point scale where 0=no pain to 100=worst pain imaginable. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-214868 3.25 μg | AGN-214868 16.25 μg | Placebo
Number analyzed (Participants) | 84 | 82 | 124
Score on a scale
  Baseline | 60.8 (22.39) | 58.4 (24.04) | 60.0 (22.39)
  Change from Baseline at Week 12 (N=82, 80, 118) | -11.7 (25.36) | -7.9 (28.61) | -11.1 (27.64)

ADVERSE EVENTS:
Description: The safety population (all participants who received at least one dose of study medication) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Groups:
- AGN-214868 3.25 μg_Cycle 1; AGN-214868 3.25 μg_ Cycle 2: One treatment of AGN-214868 injected into areas of postherpetic neuralgia pain for a total dose of 3.25 μg.
- AGN-214868 16.25 μg_Cycle 1; AGN-214868 16.25 μg_ Cycle 2: One treatment of AGN-214868 injected into areas of postherpetic neuralgia pain for a total dose of 16.25 μg.
- Placebo_Cycle 1; Placebo_Cycle 2: One treatment of Placebo to AGN-214868 injected into areas of postherpetic neuralgia pain.
Arm/Group | AGN-214868 3.25 μg_Cycle 1 | AGN-214868 16.25 μg_Cycle 1 | Placebo_Cycle 1 | AGN-214868 3.25 μg_ Cycle 2 | AGN-214868 16.25 μg_ Cycle 2 | Placebo_Cycle 2
Serious Adverse Events (participants affected / at risk) | 1/84 | 2/83 | 1/125 | 5/94 | 5/95 | 3/79
Other Adverse Events (participants affected / at risk) | 1/84 | 1/83 | 2/125 | 6/94 | 1/95 | 3/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-214868 3.25 μg_Cycle 1 (N=84) | AGN-214868 16.25 μg_Cycle 1 (N=83) | Placebo_Cycle 1 (N=125) | AGN-214868 3.25 μg_ Cycle 2 (N=94) | AGN-214868 16.25 μg_ Cycle 2 (N=95) | Placebo_Cycle 2 (N=79)
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-214868 3.25 μg_Cycle 1 (N=84) | AGN-214868 16.25 μg_Cycle 1 (N=83) | Placebo_Cycle 1 (N=125) | AGN-214868 3.25 μg_ Cycle 2 (N=94) | AGN-214868 16.25 μg_ Cycle 2 (N=95) | Placebo_Cycle 2 (N=79)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 6 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.